CLINICAL TRIAL: NCT02662543
Title: The Epidemiology and Etiology of Acute Gastroenteritis Among Estonian Children Aged < 18 Years After Introduction of Rotavirus Vaccines
Brief Title: The Epidemiology and Etiology of Acute Gastroenteritis Among Estonian Children After Introduction of Rotavirus Vaccines
Acronym: ERVS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Kadri Kõivumägi, PhD student, University of Tartu
Other Study IDs: 224/T-3
Record Dates: First submitted 2016-01-14; First posted 2016-01-25 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Rotavirus Infection
Keywords: rotavirus,; acute gastroenteritis; vaccination; Estonia; impact; severity scales
MeSH Terms: conditions — Rotavirus Infections; Tooth, Impacted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hospitalized AGE patients: Children less than 18-years-old hospitalized due to acute gastroenteritis to seven Estonian hospitals participating in this study

SUMMARY:
This study is designed to estimate the changes in the etiology and epidemiology of acute gastroenteritis in children aged less than 18 years after the implementation of rotavirus vaccine in the Estonian national immunization program in July 2014.

DETAILED DESCRIPTION:
The two-year study period started in February 2015.

The study population consists of all children less than 18-years-old hospitalized due to acute gastroenteritis (AGE) to seven Estonian hospitals participating in this study. Expected sample size is about 2000 patients.

Hospitals that participate in this study are Tartu University Hospital, West-Tallinn Central Hospital, Tallinn's Children Hospital, Pärnu Central Hospital, South-Estonian Hospital, Kuressaare Hospital and Ida-Viru Central Hospital.

Before enrollment all patients are asked to give an informed consent. After enrollment the study doctor completes electronic questionnaire regarding the patients demographic data, medical history and vaccinations. Specific database for our study has been created by company Vision 5D. After completing electronic questionnaire the doctor collects 2 stool samples each 2 ml of volume into Eppendorf tubes produced by our study laboratory. The samples are transported to our study laboratory where they are tested for rotavirus, norovirus G1, G2, astrovirus, adenovirus and sapovirus with Fast-Track Diagnostics real-time assay kit FTD Viral Gastroenteritis. The samples positive for rotavirus are refrigerated at -70 degrees for further genotyping and sequencing.

ELIGIBILITY:
Inclusion Criteria:

* children aged < 18 year
* hospitalized due to acute gastroenteritis

Exclusion Criteria:

* children aged > 18 years
* gastroenteritis due to known non-infectious causes

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children less than 18-years-old hospitalized due to acute gastroenteritis to seven Estonian hospitals participating in this study from 02.2015-09.2016
Sampling Method: Non-Probability Sample
Enrollment: 2260 (Actual)
Dates: Start 2015-02; Primary Completion 2018-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
The impact of rotavirus vaccination on hospitalizations due to acute gastroenteritis | up to 2 years
  Evaluate the impact of rotavirus vaccination on hospitalizations due to acute gastroenteritis

SECONDARY OUTCOMES:
The severity of disease according to Vesikari and Clark severity scales | up to 2 years
  Measure the severity of disease according to Vesikari and Clark severity scales

OTHER OUTCOMES:
The prevalence of rotavirus, adenovirus, astrovirus, norovirus G1, G2 and sapovirus gastroenteritis in Estonia after the implementation of rotavirus vaccine | up to 2 years
  Determine the prevalence of rotavirus, adenovirus, astrovirus, norovirus G1, G2 and sapovirus gastroenteritis in Estonia after the implementation of rotavirus vaccine
Rotavirus genotypes | up to 2 years
  Determine the genotypes of circulating rotavirus
Intussusception | up to 2 years
  Monitor the incidence of intussusception during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Irja Lutsar, PhD, Study Chair — Institute of Microbiology, University of Tartu
Locations (1):
- Department of Microbiology, University of Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koivumagi K, Soeorg H, Toompere K, Kallas E, Joegeda EL, Lass E, Huik K, Lutsar I; RV Study group. Rotavirus Strain Surveillance in Estonia After Introduction of Rotavirus Universal Mass Vaccination. Pediatr Infect Dis J. 2021 May 1;40(5):489-494. doi: 10.1097/INF.0000000000003039. PMID 33847298